CLINICAL TRIAL: NCT02351219
Title: Phase II Study of FOLFOXIRI as Primary Treatment for Stage III Unresectable Locally Advanced Pancreatic Cancer
Brief Title: FOLFOXIRI as Primary Treatment for Locally Advanced Pancreatic Cancer
Acronym: FLAP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliero, Universitaria Pisana (Other)
Responsible Party: Principal Investigator, Enrico Vasile, MD, PhD, Azienda Ospedaliero, Universitaria Pisana
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FLAP study
Record Dates: First submitted 2015-01-20; First posted 2015-01-30 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Pancreatic Carcinoma Stage III
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — FOLFOXIRI protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FOLFOXIRI (Experimental)
  Interventions: Drug: FOLFOXIRI

INTERVENTIONS:
Drug: FOLFOXIRI

SUMMARY:
The study is conducted as a monocentric prospective phase II trial. Patients with unresectable stage III locally advanced pancreatic cancer (defined for extended encasement of superior mesenteric artery/celiac axis/hepatic artery or for combined venous and arterial involvement or for unreconstructible venous encasement), ECOG PS 0-1 and age 18-75 are eligible.

After multidisciplinary evaluation of resectability, treatment with FOLFOXIRI is provided for a maximum of 12 cycles with multidisciplinary evaluation of disease status every 4 cycle.

In case of tumors have deemed resectable surgery is considered. In case tumors remain unresectable, radiotherapy is evaluated after the end of chemotherapy.

Primary objective of the study is the rate of patients who become resectable and undergo radical surgical resection after chemotherapy.

Secondary objectives are: response rate, progression-free survival, overall survival, toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Stage III unresectable pancreatic cancer defined for:

  * extended encasement of superior mesenteric artery or celiac axis/hepatic artery
  * both arterial and venous (portal vein/superior mesenteric vein) encasement
  * unreconstructible vessel encasement
* ECOG Performance Status 0-1
* Age 18-75
* Adequate liver, renal and bone marrow function

Exclusion Criteria:

* Evidence of distant metastases
* Cardiovascular diseases
* Contraindications to studied drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-12; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Radical resection rate | 6 months

SECONDARY OUTCOMES:
Progression-free survival | Within 24 months

OTHER OUTCOMES:
Overall survival | Within 36 months
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | within all the treatment period

CONTACTS AND LOCATIONS:
Locations (1):
- Azienda Ospedaliero-Universitaria Pisana, Pisa, PI, Italy